CLINICAL TRIAL: NCT05221463
Title: The Effect of Video-assisted Breastfeeding Education Given to Mothers of Hospitalized Newborns on Breastfeeding Self-efficacy and Breastfeeding Success: A Quasi-experimental Study
Brief Title: The Effect of Video-assisted Breastfeeding Education Given to Mothers of Hospitalized Newborns on Breastfeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Nazlı Baltacı, Assistant Professor, phD, Ondokuz Mayıs University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 360
Record Dates: First submitted 2022-01-22; First posted 2022-02-03 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Breastfeeding; Intensive Care Units; Neonatal
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational group (Experimental): Video-assisted breastfeeding training was given to the educational group.
  Interventions: Behavioral: Video-assisted breastfeeding training
- Control group (Other): Only the hospital's routine general breastfeeding training was given to the control group, and no other intervention was made.
  Interventions: Behavioral: The hospital's routine general breastfeeding training

INTERVENTIONS:
Behavioral: Video-assisted breastfeeding training — Breastfeeding training was given to the experimental group for 3 days by means of the training material prepared by the training nurse of the hospital about breast milk and breastfeeding and routinely used by nurses in breast milk training in neonatal units. During the training, mothers were allowed to watch breast milk and breastfeeding training videos. On the third day after the training, feedback was received from the applications in the video regarding the knowledge and skills of the mother, and the mother's questions were answered.
  Arms: Educational group
Behavioral: The hospital's routine general breastfeeding training — The control group was given the hospital's general breastfeeding training for 3 days by means of the training material prepared by the training nurse of the hospital about breast milk and breastfeeding and used routinely by nurses in breast milk training in neonatal units, and the questions of the mother were answered. The mothers in this group performed the routine breastfeeding process and no other interventions were made.
  Arms: Control group

SUMMARY:
Breastfeeding rates of infants in intensive care units in the world and in Turkey are undesirably low due to the conditions of infants, mothers and healthcare workers, which threatens the health of newborns in many aspects in the early and future periods. It is thought that the visual materials and tools used in breastfeeding education can be effective both in the permanence of the acquired knowledge and in the transformation of the knowledge into behavior. This study was conducted to determine the effect of video-assisted breastfeeding and breastfeeding education given to mothers of hospitalized newborns on breastfeeding self-efficacy and breastfeeding success.

Hypotheses Hypothesis 01: Video-assisted breastfeeding and breastfeeding education given to mothers of hospitalized newborns does not affect breastfeeding self-efficacy of mothers.

Hypothesis 1: Video-assisted breastfeeding and breastfeeding education given to mothers of hospitalized newborns increases mothers' breastfeeding self-efficacy.

Hypothesis 02: Video-assisted breast milk and breastfeeding education given to mothers of hospitalized newborns does not affect mothers' breastfeeding success.

Hypothesis 2: Video-assisted breastfeeding and breastfeeding education given to mothers of hospitalized newborns increases the breastfeeding success of mothers.

This research is a non-randomized quasi-experimental study in a two-group pretest-posttest design. The research was carried out in the neonatal intensive care level 2 unit of a university hospital located in the north of Turkey. In the study, mothers who met the inclusion criteria were assigned to the education group (EG) (n=44) and the control group (CG) (n=44), some mothers did not continue the education program and left the study. In this case, the study was completed with 41 mothers in EG and 43 mothers in CG. Video assisted breastfeeding training was given to the intervention group. Only the hospital's routine general breastfeeding training was given to the control group, and no other intervention was made.Breastfeeding self-efficacy with the Postpartum Breastfeeding Self-Efficacy Scale-Short Form and breastfeeding success levels with the LATCH Breastfeeding Diagnostic Measurement Tool were evaluated at the beginning of the study (pretest) and after three days of breastfeeding training (posttest).

DETAILED DESCRIPTION:
Breastfeeding rates of infants in intensive care units in the world and in Turkey are undesirably low due to the conditions of infants, mothers and healthcare workers, which threatens the health of newborns in many aspects in the early and future periods. The education given to the mother by health care professionals; It has a great effect on the initiation and maintenance of breastfeeding, prevention of breast complications and successful breastfeeding. It is thought that the visual materials and tools used in breastfeeding education can be effective both in the permanence of the acquired knowledge and in the transformation of the knowledge into behavior. This study was conducted to determine the effect of video-assisted breastfeeding and breastfeeding education given to mothers of hospitalized newborns on breastfeeding self-efficacy and breastfeeding success.

This research is a non-randomized quasi-experimental study in a two-group pretest-posttest design. The research was carried out in the neonatal intensive care level 2 unit of a university hospital located in the north of Turkey.

The universe of the study consisted of mothers who were hospitalized in the neonatal intensive care unit of the hospital where the study was conducted between 01.06.2021 and 25.12.2021 and came to breastfeed. Power analysis was performed using the G*Power (v3.1.7) program to determine the number of samples.In the calculation made by assuming that the evaluations to be made between two independent groups will have a large effect (d=0.80) on the Breastfeeding Self-Efficacy Scale-Short Shape scale scores (Tokat et al. 2010), in order to obtain 80% power (1-β) at the α=0.05 level. It was determined that there should be at least 36 people in each group. Considering that there may be losses during the research process, it was planned to recruit 44 people to each group. Three of the mothers (n=44) who met the inclusion criteria and were included in the training group (EG), and one of the mothers (n=44) who were included in the control group (KG) dropped out of the study by not continuing the training program. In this case, the study was completed with 41 mothers in EG and 43 mothers in CG.

The suitability of the mothers who came to the neonatal intensive care unit to breastfeed their babies was evaluated by the researcher. The mothers who were willing and able to participate in the study were given the necessary information about the study and their written consent was obtained. The study had an intervention and a control group. The researcher first gave video-assisted breastfeeding training to the intervention group for 3 days. On the third day after the training, feedback was received from the applications in the video regarding the knowledge and skills of the mother, and the mother's questions were answered. When these trainings were completed, other eligible mothers were included in the control group. The control group was given only the hospital's routine general breastfeeding training for 3 days and the questions of the mother were answered. The mothers in this group performed the routine breastfeeding process and no other interventions were made.

First of all, sociodemographic and obstetric data of the mothers were collected by using the introductory information form, and information about the infants was obtained by the researcher from the infants' files. Breastfeeding self-efficacy with the Postpartum Breastfeeding Self-Efficacy Scale-Short Form and breastfeeding success levels with the LATCH Breastfeeding Diagnostic Measurement Tool were evaluated at the beginning of the study (pretest) and after three days of breastfeeding training (posttest) before the training was given.

Before starting this study, ethics committee approval was obtained from the Clinical Research Ethics Committee of a University in northern Turkey (decision dated 28/05/2021, numbered 2021/239) and written permission from the relevant institution where the study was conducted. In addition, the purpose of the study was explained to all participants before the data collection form was applied, and written informed consent was obtained from those who volunteered to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* wanting to participate
* healthy
* 18 years and older
* the baby is hospitalized and breastfed by the neonatologist is deemed appropriate
* able to read and write
* no psychiatric problems
* mothers who speak Turkish

Exclusion Criteria:

* unwilling to participate
* patient
* breast-feeding not approved by the neonatologist
* having breast problems that prevent breastfeeding
* mental, cognitive, psychiatric, hearing and vision problems
* illiterate
* mothers who do not speak Turkish

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-25 (Actual); Study Completion 2021-12-25 (Actual)

PRIMARY OUTCOMES:
Breastfeeding self-efficacy change | At baseline and at the end of the 3nd day of study, breastfeeding self-efficacy was assessed
  As assessed by the Postpartum Breastfeeding Self-Efficacy Scale-Brief Form.The scale assesses how competent mothers feel about breastfeeding. The lowest score that can be obtained from the scale is 14, and the highest score is 70. The higher the score, the higher the breastfeeding self-efficacy.
Breastfeeding success change | At baseline and at the end of the 3nd day of study, breastfeeding success was assessed
  As assessed by the LATCH (Latch on breast, Audible swallowing, Type of nipple, Comfort bresat/nipple, Hold) Breastfeeding Diagnostic Measurement Tool. The scale consists of five evaluation criteria [L (Latch on the breast), A (Audible swallowing), T (Type of the nipple), C (Comfort breast/nipple), H (Hold)]. Each item is evaluated between 0 and 2 points. A maximum of 10 points can be obtained from the scale. As the score obtained from the scale increases, the success of breastfeeding increases.

CONTACTS AND LOCATIONS:
Overall Officials: Nazlı Baltacı, phD, Principal Investigator — Ondokuz Mayıs University; Esra Tural Büyük, phD, Principal Investigator — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayıs University Health, Application and Research Center, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available from the corresponding author (E.T.B.) upon reasonable request.